CLINICAL TRIAL: NCT04501302
Title: Effect of Four Abdominal and Pelvic Exercises on the Inter-recti Distance in Women: an Observational Study
Brief Title: Effect of Four Exercises on the Inter-recti Distance in Women
Acronym: Traecho
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: APOR B de Gasquet (Other)
Responsible Party: Sponsor
Other Study IDs: TrAEcho01
Record Dates: First submitted 2020-07-09; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Diastasis, Muscle
Keywords: transversus abdominis, diastasis rectus abdominis, exercise, pelvic floor muscles
MeSH Terms: conditions — Diastasis, Muscle; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diastasis rectus abdominis (DRA) is defined as an excessive separation between the two abdominal rectus muscles. It is generally quantified by the inter-recti distance. In postpartum women, the prevalence of diastasis is 60% six weeks after delivery.

The increase in the inter-recti distance has been associated with a decrease in strength and endurance of the trunk flexors and rotators (p < 0.05). Exercise during pregnancy has been shown to be helpful in the treatment of DRA. Nevertheless, there is still not strong evidence to establish what kind of exercise should be recommended during pregnancy and in postpartum.

The aim of this study is to compare the morphological and functional changes of the linea alba during four exercises.

Inter-recti distance, linea alba thickness and distortion index will be measured at rest, as well as during 4 exercises (draw in maneuver, crunch, pelvic floor muscle contraction and a "de Gasquet" exercise). Subgroup analysis will be performed to determine if the presence or absence of an abdominal diastasis has an influence on these outcomes.

A cross-sectional pilot study will be carried out. The main outcome measure will the inter-recti distance. Secondary outcomes will be the thickness of linea alba and distortion index.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Parous
* Women
* Accepting to participe in the research

Exclusion Criteria:

* Under curatorship
* Persons deprived of their liberty by judicial or administrative decision
* Having intellectual limitations that may limit the understanding of questionnaires or exercises
* With limitations in understanding the French language
* Pregnant women
* History of pelvic / spine fractures
* History of pelvic surgery
* History of spinal surgery
* History of abdominal surgery
* History of lower limbs weakness, changes in osteotendinous reflexes or loss of sensitivity

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult parous women attending to several physiotherapy centers in Paris will be recruited
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2020-09-25 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Inter-recti distance | During the exercise
  The distance between the two medial borders of rectus abdominis muscles is measured using ultrasound

SECONDARY OUTCOMES:
Linea alba thickness | During the exercise
  Linea alba thickness is measured using ultrasound
Distortion index of the linea alba | During the exercise
  Average deviation of the linea alba from the shortest path between the recti measured using ultrasound

OTHER OUTCOMES:
Transversus abdominis thickness | During the exercise
  Transversus abdominis thickness at 1cm lateral from the fascia transversalis measured using ultrasound
Current lumbopelvic pain intensity | During the assessement
  Current lumbopelvic pain will be measured using a visual analog scale
Acute lumbopelvic pain severity | During the assessement
  The participants will be asked about their lumbopelvic pain mean intensity in the last week using a visual analog scale
Chronic lumbopelvic pain severity | During the assessement
  The participants will be asked about their lumbopelvic pain mean intensity in the last 6 months using a visual analog scale
Urinary symptoms | During the assessement
  Urinary symptoms will be measured using the Urinary Symptom Profile questionnaires

IPD SHARING:
Plan to Share IPD: Undecided